CLINICAL TRIAL: NCT04464902
Title: The Effects of Knee Extension Constraint Rehabilitation After ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR001
Record Dates: First submitted 2020-06-30; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; injury prevention; knee extension constraint
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients and investigator all don't know which group they participated in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- knee extension constraint rehabilitation group (Other)
  Interventions: Device: brace1
- placebo group (Other)
  Interventions: Device: brace2
- control group (Other)
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: brace1 — The brace1 can provide resistance when patients want to extend their knee.
  Arms: knee extension constraint rehabilitation group
Device: brace2 — The brace1 can't provide resistance when patients want to extend their knee.
  Arms: placebo group
Other: No Intervention — Control Group don't have any brace.
  Arms: control group

SUMMARY:
To develop new prevention programs for non-contact ACL injuries that do not require additional training time and assistance from a sports medicine professional personnel. A knee extension constraint will be utilized to patients who have undertaken ACL reconstruction.

And to determine the effects of knee extension constraint rehabilitation on lower extremity biomechanics after ACL reconstruction surgery.

DETAILED DESCRIPTION:
Purpose Of exploring the biomechanical effect of knee extension constraint rehabilitation on rehabilitation after anterior cruciate ligament (ACL) reconstruction. Methods: Recruit 60 patients after ACL reconstruction. Divide them into three groups by random block method: Knee extension constraint rehabilitation group (wearing a brace with limitation of knee extension), Placebo group (wearing a brace without limitation of knee extension), and Control group (no brace is worn). The three groups of patients received the same rehabilitation training from 1 to 12 weeks after surgery, starting from week 13 and intervening on the first day of each week (wearing braces). Five tests were performed at the end of the 12th, 24th, 36th, and 48th weeks after surgery. Vicon system and force platform system will be synchronized used to test walking, jogging, side-cutting, and jumping; The Isokinetic dynamometer system will be used to test muscle strength. Outcome evaluation indicators and statistical methods: (1) Mixed design two-way analysis of variances will be used for the following indicators: approach run velocity and jump height; knee flexion angle at initial foot contact with the ground; knee extension moment at the time of peak impact poster ground reaction force, study group will be considered as an independent variable while testing time as the variable for repeated measurements. (2) The knee flexion, valgus-varus, and internal-external rotation angles, and extension, valgus-varus, and internal-external rotation moments of each leg during support phase of each movement will be expressed as functions of normalized movement time and leg (involved or uninvolved) using regression analysis with dummy variable. A dummy variable will be used to represent involved and uninvolved legs. A forward elimination procedure will be used to determine the best regression equations. The regression procedure will be stopped when the contributions of powers of n+1 and n+2 have no significant contribution to the overall regression. The contribution of the dummy variable in the regression will be an indication of asymmetry of the movements of involved and uninvolved legs. The effect of study group on movement asymmetry will be determined by comparing the contribution of dummy variables to the overall regression among study groups using a one-way ANOVA. The effects of study group and testing time on the ACL injury risk index will be determined for each knee in each movement using two-way ANOVA with mixed model. Study group will be considered as an independent variable while testing time as a repeated measure variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have isolated ACL injury and receive ACL reconstruction surgery at Sports Medicine Center, 3rd Hospital of Beijing University, Beijing, China.
* 18-35 years old
* With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures).
* All participants have no known disorders or diseases other than ACL rupture.

Exclusion Criteria:

* Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07-28 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
walking speed | at 24 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
walking speed | at 36 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
walking speed | at 48 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
ground reaction force | at 24 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
ground reaction force | at 36 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
ground reaction force | at 48 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
knee flexion angle | at 24 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
knee flexion angle | at 36 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
knee flexion angle | at 48 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | at 24 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | at 36 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | at 48 weeks after ACL reconstruction surgery.
  Three-dimensional gait analysis system were used during walking, jogging, cutting and jumping.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | at 24 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
The International Knee Documentation Committee (IKDC) score | at 36 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.
The International Knee Documentation Committee (IKDC) score | at 48 weeks after ACL reconstruction surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No